CLINICAL TRIAL: NCT06268340
Title: Preservation of Hearing and Structure Using an Electrocochleography Based Corrective Action Guide
Brief Title: Hearing and Structure Preservation Via ECochG
Acronym: PRESERVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABIntl-23-25
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss, Sensorineural; Severe-to-profound Hearing Loss
Keywords: Electrocochleography; Hearing Preservation; Structure Preservation; Intra-cochlear monitoring; Scalar translocations; Cochlear Microphonics; Corrective action guide; Cochlear Implants
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): ECochG monitored CI surgery incl. corrective action guide
  Interventions: Procedure: ECochG monitored CI surgery incl. corrective action guide
- Control (Active Comparator): Routine CI surgery without ECochG monitoring
  Interventions: Procedure: Routine CI surgery without ECochG monitoring

INTERVENTIONS:
Procedure: ECochG monitored CI surgery incl. corrective action guide — Interventional surgery with surgeon having access to intra-operative ECochG monitoring feedback to deploy ECochG based corrective action guide
  Arms: Intervention
Procedure: Routine CI surgery without ECochG monitoring — Routine CI surgery with access to ECochG monitoring by surgeon
  Arms: Control

SUMMARY:
The goal of the study is to determine the benefit of using an ECochG-based corrective action guide during cochlear implant surgery compared to the traditional surgical approach without ECochG surveillance and guidance.

DETAILED DESCRIPTION:
Cochlear implantation is a highly effective method of rehabilitating hearing in individuals with severe to profound hearing loss. One current hurdle to optimising hearing outcomes following cochlear implantation is the unavoidable trauma caused to the inner ear during implant surgery. This damage can mean residual hearing that would remain valuable following implantation is lost. Various approaches have been trialed to preserve hearing during implantation surgery, modifying implantation technique and administering steroids. Electrocochleography (ECochG) is a monitoring technique that can be used during electrode insertion to record inner ear structural integrity and function.

The PRESERVE trial is an international, multi-centre, randomised controlled trial. The trial will randomly allocate adult cochlear implant recipients to undergo implantation surgery either with ECochG-guidance, or via the standard approach without guidance. Participants will be blinded, meaning they will not know which group they will be allocated to. Where ECochG is used, evidence of damage during insertion detected with the monitoring will trigger the surgeon to follow a corrective pathway. All other aspects of surgery and post operative care will follow standard clinical pathways for both groups.

Participants will have their natural hearing measured preoperatively, and 3- and 6-months following implant activation. The change in natural hearing thresholds at different frequencies, and the degree of hearing preservation will then be calculated and compared between the standard surgery and ECochG-guided group. Using their cochlear implant, understanding of speech will also be measured and compared between groups. In addition, participants will undergo a second CT scan following implantation surgery, and this will be compared to the routine pre-operative imaging to assess both the location of the implant electrode, and structural preservation of the cochlear. Throughout the study participants will remain under the care of their routine medical team.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or older
* Within cochlear implant inclusion criteria by local regulations/guidelines at the time of implantation
* Severe to profound hearing loss (average air conduction unaided hearing threshold of ≥ 70 dB HL for 500, 1000, 2000 and 4000 Hz) in the ear to be implanted
* Air conduction unaided hearing threshold ≤ 70 dB HL at 500 Hz in the ear to be implanted
* Less than 15 years of severe to profound deafness on the implant ear prior to surgery
* Post-lingually acquired hearing loss in the ear to be implanted
* Normal cochlear anatomy as confirmed by pre-operative imaging in the ear to be implanted
* Listed for an Advanced Bionics HiRes Ultra (3D) HiFocus SlimJ electrode array
* Listed for cochlear implant surgery under general anaesthesia
* Fluent in local language
* Given informed consent to participate in the study

Exclusion Criteria:

* Abnormal cochlear anatomy (including ossification) as identified by pre-operative radiological evaluation in the ear to be implanted
* Any pre-existing cochlear or middle ear pathology, such as otosclerosis, cholesteatoma, or previous middle ear surgery in the ear to be implanted
* Any medical conditions that would increase the risk of local complications during cochlear implantation, such as autoimmune diseases or active local infections
* Diagnosis of auditory spectrum neuropathy disorder
* Deafness due to lesions of the acoustic nerve or central auditory pathway
* Deafened by meningitis
* Single sided deafness (average for 500, 1000, 2000 and 4000 Hz in the better ear ≤ 30 dB HL)
* Asymmetric hearing loss (average for 500, 1000, 2000 and 4000 Hz in the better ear > 30 dB HL and ≤ 55 dB HL)
* History of previous cochlear implantation/re-implantation on either ear
* Any contraindications to computed tomography (CT) scans
* Concurrent participation in other cochlear implant related studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hearing Preservation | From pre-operative to 6 months post-operative
  Difference in dB (absolute) and % (relative) in low-frequency hearing preservation measured via air conduction pure tone audiometry

SECONDARY OUTCOMES:
Structure Preservation | 1 month post-operative
  Difference in mm of structure preservation (distance from electrode contact to basilar membrane) via radiological assessment of the position of the electrode array
Speech perception | From pre-operative to 6 months post-operative
  Difference in speech perception scores in both quiet (%) and noise (dB SNR) using the International Matrix Test

OTHER OUTCOMES:
Surgeons' feedback | Through study completion, an average of 2.5 years
  Qualitative feedback on surgical experience measured via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Matt E Smith, Dr, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (7):
- Universitair Ziekenhuis Gent, Ghent, Gent, Belgium
- Le Centre Hospitalier Régional Universitaire de Tours, Tours, Tours, France
- Universitätsklinikum Freiburg Klinik, Freiburg im Breisgau, Freiburg, Germany
- Ospedale Martini, Torino, TO, Italy
- World Hearing Center, Warsaw, Nadarzyn, Poland
- Hospital Universitario Clinico San Cecilio, Granada, Granada, Spain
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bester C, Collins A, Razmovski T, Weder S, Briggs RJ, Wei B, Zakaria AF, Gerard JM, Mitchell-Innes A, Tykocinski M, Kennedy R, Iseli C, Dahm M, Ellul S, O'Leary S. Electrocochleography triggered intervention successfully preserves residual hearing during cochlear implantation: Results of a randomised clinical trial. Hear Res. 2022 Dec;426:108353. doi: 10.1016/j.heares.2021.108353. Epub 2021 Sep 20. PMID 34600798
- [Background] Buechner A, Bardt M, Haumann S, Geissler G, Salcher R, Lenarz T. Clinical experiences with intraoperative electrocochleography in cochlear implant recipients and its potential to reduce insertion trauma and improve postoperative hearing preservation. PLoS One. 2022 Apr 22;17(4):e0266077. doi: 10.1371/journal.pone.0266077. eCollection 2022. PMID 35452461
- [Background] Carlson ML, Driscoll CL, Gifford RH, Service GJ, Tombers NM, Hughes-Borst BJ, Neff BA, Beatty CW. Implications of minimizing trauma during conventional cochlear implantation. Otol Neurotol. 2011 Aug;32(6):962-8. doi: 10.1097/MAO.0b013e3182204526. PMID 21659922
- [Background] Dalbert A, Sim JH, Gerig R, Pfiffner F, Roosli C, Huber A. Correlation of Electrophysiological Properties and Hearing Preservation in Cochlear Implant Patients. Otol Neurotol. 2015 Aug;36(7):1172-80. doi: 10.1097/MAO.0000000000000768. PMID 25839980
- [Background] Moore FL, Miller LJ. Stress-induced inhibition of sexual behavior: corticosterone inhibits courtship behaviors of a male amphibian (Taricha granulosa). Horm Behav. 1984 Dec;18(4):400-10. doi: 10.1016/0018-506x(84)90026-6. PMID 6097527
- [Background] Blackford HN, Murray K, Stephenson TP, Mundy AR. Results of transvesical infiltration of the pelvic plexuses with phenol in 116 patients. Br J Urol. 1984 Dec;56(6):647-9. doi: 10.1111/j.1464-410x.1984.tb06137.x. PMID 6534483
- [Background] Gifford RH, Dorman MF, Skarzynski H, Lorens A, Polak M, Driscoll CL, Roland P, Buchman CA. Cochlear implantation with hearing preservation yields significant benefit for speech recognition in complex listening environments. Ear Hear. 2013 Jul-Aug;34(4):413-25. doi: 10.1097/AUD.0b013e31827e8163. PMID 23446225
- [Background] Lenarz T, Timm ME, Salcher R, Buchner A. Individual Hearing Preservation Cochlear Implantation Using the Concept of Partial Insertion. Otol Neurotol. 2019 Mar;40(3):e326-e335. doi: 10.1097/MAO.0000000000002127. PMID 30741914
- [Background] O'Leary S, Mylanus E, Venail F, Lenarz T, Birman C, Di Lella F, Roland JT Jr, Gantz B, Beynon A, Sicard M, Buechner A, Lai WK, Boccio C, Choudhury B, Tejani VD, Plant K, English R, Arts R, Bester C. Monitoring Cochlear Health With Intracochlear Electrocochleography During Cochlear Implantation: Findings From an International Clinical Investigation. Ear Hear. 2023 Mar-Apr 01;44(2):358-370. doi: 10.1097/AUD.0000000000001288. Epub 2022 Nov 8. PMID 36395515
- [Background] Saoji AA, Patel NS, Carlson ML, Neff BA, Koka K, Tarigoppula VSA, Driscoll CLW. Multi-frequency Electrocochleography Measurements can be Used to Monitor and Optimize Electrode Placement During Cochlear Implant Surgery. Otol Neurotol. 2019 Dec;40(10):1287-1291. doi: 10.1097/MAO.0000000000002406. PMID 31644474
- [Background] Brown DC, Conzemius MG, Shofer F, Swann H. Epidemiologic evaluation of postoperative wound infections in dogs and cats. J Am Vet Med Assoc. 1997 May 1;210(9):1302-6. PMID 9143534
- [Background] Verberne J, Risi F, Campbell L, Chambers S, O'Leary S. The Effect of Scala Tympani Morphology on Basilar Membrane Contact With a Straight Electrode Array: A Human Temporal Bone Study. Otol Neurotol. 2017 Jan;38(1):47-53. doi: 10.1097/MAO.0000000000001259. PMID 27755369
- See also: Cochlear implants for children and adults with severe to profound deafness - Technology appraisal guidance [TA566] — https://www.nice.org.uk/guidance/ta566